CLINICAL TRIAL: NCT06246929
Title: Comorbidity of Chronic Pain and Early Cognitive Decline Among Older, Community-Based Black Adults: Comparative Effectiveness of Mindfulness-Based Cognitive Therapy With Walking (MBCT+w) vs Active Living Every Day (ALED)
Brief Title: Healthy Aging as Black Adults, In It Together: a Comparative Effectiveness Study of Chronic Pain and Cognitive Decline
Acronym: HABIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Olivia I.Okereke, MD, Director of Geriatric Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000002
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Physical Activity; Older Adults; Mild Cognitive Impairment
Keywords: Black Older Adults; African Americans; Subjective Cognitive Decline; Memory Related Problems; Pain; Cognition Disorders
MeSH Terms: conditions — Chronic Pain; Motor Activity; Cognitive Dysfunction; Pain; Cognition Disorders

STUDY DESIGN:
Masking Description: Study Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy With Walking (MBCT+w) (Experimental): MBCT+w uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions and weekly practice assignments (homework). The MBCT+w sessions teach skills and strategies to manage early cognitive concerns and chronic pain. The format is an 8-week program with 90-minute weekly meetings that will focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. MBCT+w uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Interventions: Behavioral: MBCT+w
- Active Living Every Day (ALED) (Active Comparator): ALED is a behavior change program. ALED offers different options to traditional exercise program to help participants overcome barriers to physical activity and increase their physical activity. The format is a 12-week program with 60-minute sessions that include a short lecture and group discussions to help participants set goals, decrease barriers to exercise, and find an activity they enjoy. The ALED program is conducted in the same format as MBCT+w, but participants are not taught the mind-body, walking or cognitive-behavioral skills. ALED will also use a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Interventions: Behavioral: ALED

INTERVENTIONS:
Behavioral: MBCT+w — MBCT+w uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions and weekly practice assignments (homework). The MBCT+w sessions teach skills and strategies to manage early cognitive concerns and chronic pain. The format is an 8-week program with 90-minute weekly meetings that will focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. MBCT+w uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Arms: Mindfulness-Based Cognitive Therapy With Walking (MBCT+w)
Behavioral: ALED — ALED is a behavior change program. ALED offers different options to traditional exercise program to help participants overcome barriers to physical activity and increase their physical activity. The format is a 12-week program with 60-minute sessions that include a short lecture and group discussions to help participants set goals, decrease barriers to exercise, and find an activity they enjoy. The ALED program is conducted in the same format as MBCT+w, but participants are not taught the mind-body, walking or cognitive-behavioral skills. ALED will also use a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Arms: Active Living Every Day (ALED)

SUMMARY:
The investigators aim to conduct a randomized controlled trial to compare two symptom-management programs for Black older adults with early cognitive decline (self-reported confirmed by testing) and chronic pain. The programs are Mindfulness-Based Cognitive Therapy with Walking (MBCT+w) and Active Living Every Day (ALED). The investigators will assess how each program may help in improving physical, cognitive, and emotional function. The investigators will also assess whether improvements in outcomes from the two programs are maintained through a 6-month follow-up.

DETAILED DESCRIPTION:
The investigators aim to conduct a randomized controlled trial to compare two symptom-management programs for Black older adults with early cognitive decline (self-reported or confirmed by testing) and chronic pain. The programs are Mindfulness-Based Cognitive Therapy with Walking (MBCT+w) and Active Living Every Day (ALED). The investigators will assess how each program may help in improving physical, cognitive, and emotional function outcomes. The investigators will also assess whether improvements in outcomes from the two programs are maintained through a 6-month follow-up.

The program MBCT+w is focused on learning about managing chronic pain and early cognitive decline and strategies to become more active. The ALED program focuses on learning and understanding the process of successful lifestyle change, incorporating physical activity in your day-to-day life, and strategies to manage daily activity.

The MBCT+w group meets in person for eight sessions for 90-minutes, and the ALED group meets in person for twelve sessions for 60-minutes. Each group has up to 10-12 participants. Participants receive a treatment manual. The investigators will assess how each program may help in improving physical, cognitive, and emotional function outcomes. Outcomes will be assessed at 3 points: baseline, post program, and 6-month follow-up. Assessments involve self-report questionnaires, a walk test, and a neuropsychological exam. The investigators will assess whether improvements in outcomes from the two programs are maintained through a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Black adults, male and females, age 50 or older
* Have nonmalignant musculoskeletal chronic pain for more than three months
* Reports early cognitive decline (subjective and objective)
* Telephone Interview for Cognitive Status-41 score greater than or equal to 31
* Functional Activities Questionnaire score less than 9
* English fluency/literacy
* Free of concurrent psychotropic or pain medication for at least 2 weeks prior to initiation of treatment, OR stable on current psychotropic or pain medication for a minimum of 6 weeks and willing to maintain stable dose
* Cleared by medical doctor for study participation and no self-reported concerns about physical functioning on the revised Physical Activity Readiness Questionnaire (PAR-Q; score 0)

Exclusion Criteria:

* Diagnosed with dementia or neurodegenerative disease
* Regular use of nonpharmacological pain management
* Diagnosed with serious mental illness or substance abuse
* Current suicidal ideation on self-report
* Engagement of regular exercise for more than 30 minutes daily
* Unable to walk

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function | 0 Weeks, 12 Weeks, 6 Months
  Change in participant's self-reported performance of everyday physical activities, with items ranging from 1-4. Higher T scores indicate greater physical function.

SECONDARY OUTCOMES:
ActiGraph GT9X Link Accelerometer | 0 Weeks, 12 Weeks, 6 Months
  Measure the change in steps during the 7 days preceding baseline assessment, throughout intervention period, and 7 days preceding 6-month follow-up.
Six-minute walk test (6MWT) | 0 Weeks, 12 Weeks, 6 Months
  Assesses distance walked in 6 minutes.
Montreal Cognitive Assessment (MoCA) | 0 Weeks, 12 Weeks, 6 Months
  A comprehensive test that assesses eight cognitive abilities (orientation, short-term memory, executive function, clock drawing, animal naming, language abilities, abstraction, and attention). Higher total scores (0-30) indicate greater cognitive functioning.
Everyday Cognitive Scale (eCog-12) | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported cognitively mediated functional abilities, with items ranging 1-5. Scores are calculated by averaging the 12 items, and range 1-5, with higher scores indicating greater cognitive decline.
PROMIS Depression | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported negative mood, social cognition and views of self, with items ranging from 1-5. Higher T scores indicate high levels of depression.
PROMIS Anxiety | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported fear, anxious, hyperarousal and somatic symptoms pertaining to arousal, with items ranging from 1-5. Higher T scores indicate higher levels of anxiety.

OTHER OUTCOMES:
Numerical Rating Scale (NRS) | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported pain at rest and with activity using a Likert Scale with 0 being no pain and 10 being worst possible pain.
UCLA loneliness scale 8-item (UCLA-8) | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported subjective feelings of loneliness and social isolation, with items ranging 0-3. Higher scores indicate higher feelings of loneliness.
PROMIS Emotional Support v4a | 0 Weeks, 12 Weeks, 6 Months
  Rating of participant's self-reported subjective feelings of emotional support from others, with items ranging 1-5. Higher T scores indicate higher emotional support.
Zarit Burden Interview (12-item) | 0 Weeks, 12 Weeks, 6 Months
  Rating of caregiver's self-reported subjective feelings of his or her levels of burden for caring for a person with a particular diagnosis, with items ranging 0-4. Higher scores indicate greater feelings of burden.
Caregiver Strain Questionnaire Short Form | 0 Weeks, 12 Weeks, 6 Months
  Rating of caregiver's self-reported subjective feelings of strain experienced with sleep, finances, physical movements, and emotional adjustments, with items ranging 0-1. Higher scores indicate greater feelings of strain.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Okereke, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mace RA, Gates MV, Popok PJ, Kulich R, Quiroz YT, Vranceanu AM. Feasibility Trial of a Mind-Body Activity Pain Management Program for Older Adults With Cognitive Decline. Gerontologist. 2021 Nov 15;61(8):1326-1337. doi: 10.1093/geront/gnaa179. PMID 33159516
- [Background] Mace RA, Gates MV, Bullard B, Lester EG, Silverman IH, Quiroz YT, Vranceanu AM. Development of a Novel Mind-Body Activity and Pain Management Program for Older Adults With Cognitive Decline. Gerontologist. 2021 Apr 3;61(3):449-459. doi: 10.1093/geront/gnaa084. PMID 32601670